CLINICAL TRIAL: NCT06127420
Title: Comprehensive Assessment on Diagnostic and Prognostic Performance of Coronary Physiological Indices in Patients Referred to Angiography
Brief Title: Comprehensive Assessment on Diagnostic and Prognostic Performance of Coronary Physiological Indices
Acronym: CONCORDE
Status: Active, not recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Junbo Ge, Professor, Shanghai Zhongshan Hospital
Other Study IDs: ZSCD2023001
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patients: All patients referred to angiography and undergo assessment with coronary pressure sensor
  Interventions: Other: coronary physiological indices

INTERVENTIONS:
Other: coronary physiological indices — Resting distal coronary to aortic pressure ratio, Fractional flow reserve, Resting full-cycle ratio, Coronary Flow Reserve, Microvascular resistance

SUMMARY:
The objective of the Zhongshan Hospital CONCORDE Registry is to evaluate utility, diagnostic value, and clinical outcomes of coronary physiological indices in an all-comers population of patients with suspected coronary artery disease referred to invasive coronary angiography in order to further inform patients and health care providers about which technologies are most effective and efficient in the diagnosis and management of coronary artery diseases.

DETAILED DESCRIPTION:
CONCORDE registry offers a comprehensive pressure and/or flow measurements, as well as angiography-derived functional assessment of coronary. Patient treatment was at the operator's discretion at the time of the invasive procedure. A standardized data collection sheet was used and data were extracted from electrical medical history according to standardized definition of patient's baseline characteristics, clinical outcomes, and physiologic data.

ELIGIBILITY:
Inclusion Criteria:

* suspected coronary artery disease
* referred to invasive coronary angiography

Exclusion Criteria:

* hemodynamic instability

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A all-comer population of patients with suspected coronary artery disease referred to invasive angiography at Zhongshan Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac events (MACE) | 5 years
  Cumulative incidence of a composite of any death, any myocardial infarction, or any ischemia-driven revascularization

SECONDARY OUTCOMES:
Target vessel failure (TVF) | 5 years
  Cumulative incidence of a composite of cardiac death, target-vessel related myocardial infarction, or target-vessel revascularization
Individual components of MACE and TVF | 5 years
  Cumulative incidence of the individual components of MACE and TVF

CONTACTS AND LOCATIONS:
Overall Officials: Chenguang Li, Study Director — Shanghai Zhongshan Hospital
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No